CLINICAL TRIAL: NCT00284882
Title: The Epidemiology of Group A Streptococcal Infections in Fiji (Fiji GrASP) Part 3: The Incidence of Group A Streptococcal Pharyngitis and the Prevalence of Pyoderma and Scabies in School Children in Fiji, and Establishing Immunologic Correlates of Protection for a J8 Vaccine
Brief Title: Incidence of Group A Strep Pharyngitis in School Children in Fiji
Status: Completed | Type: Observational
Sponsor: National Institute of Allergy and Infectious Diseases (NIAID) (NIH)
Other Study IDs: 05-0117
Record Dates: First submitted 2006-01-30; First posted 2006-02-01 (Estimated); Last update posted 2008-01-25 (Estimated); Status verified 2007-10

CONDITIONS: Streptococcus Group A
Keywords: Streptococcus, Fiji, pyoderma, pharyngitis, scabies
MeSH Terms: conditions — Pyoderma; Pharyngitis; Scabies

STUDY DESIGN:
Time Perspective: Prospective

SUMMARY:
The purpose of this study is to find out how often group A Streptococcus (GAS) occurs in school-age children of Central Fiji. This bacterium often causes pharyngitis (sore throat) and can also cause pyoderma (skin infection) or scabies. Approximately 1000 children ages 5-14 years will be enrolled from 4 primary schools in Central Fiji. These children will have throat swabs performed to determine how commonly GAS occurs. Over the next 10 months, children in this group who complain of sore throat will be examined and have throat swabs to determine if GAS is the cause. A subset of 600 children will be examined for pyoderma and scabies and have throat swabs every 2 months during the 10 month study. In addition, a small amount of blood will be drawn at 0, 6, and 10 months to determine the level of antibodies to Streptococcus.

DETAILED DESCRIPTION:
This study is the third part of a series of 5 studies including DMID protocols 05-0081, 05-0082, 05-0118, and 06-0081. The primary objectives of this prospective cohort study are to estimate the incidence of group A streptococcal (GAS) pharyngitis in 1000 primary school aged school children in Fiji and to assess titers of anti-J8 antibodies and correlate titers of these antibodies against GAS infection in 600 primary school aged children in Fiji. Secondary objectives are to: estimate the point prevalence of GAS pyoderma in 600 primary school aged children in Fiji; estimate the point prevalence of scabies in 600 primary school aged children in Fiji; determine the pharyngeal carriage rate of group A streptococci in 1000 primary school aged children in Fiji; describe the clinical features of GAS pharyngitis in 1000 primary school aged children in Fiji; determine the upper limit of normal values for streptococcal serology (antistreptinolysin O and anti-DNase B); genotypically characterize group A streptococci isolated from throat swabs from primary school aged children with pharyngitis; genotypically characterize group A streptococci isolated from skin swabs from pyoderma lesions in school aged children in Fiji; and determine antimicrobial susceptibility to penicillin, clindamycin, erythromycin and chloramphenicol in 150 GAS isolates from skin swabs and 150 GAS isolates from throat swabs. Approximately 1000 school children aged 5 -14 from 4 primary schools will be enrolled in the study with approximately 600 of these 1000 school children aged 5-14 from 3 of the schools in the substudy. Children in the main study will participate for 1-2 days, and children in the substudy will participate for a 10-month period. All children at the start of the study will have swabs taken to determine the pharyngeal carriage rate of GAS. Over the next 10 months school children will be examined for pharyngitis when they complain of sore throat and throat swabs will be taken to prove GAS as the etiology of clinical pharyngitis. In a subset of 600 children, sera will be taken at 0, 6 and 10 months. Skin will be examined for pyoderma and scabies and swabs will be taken from pyoderma lesions every 2 months for 10 months. Streptococcal serology, antistreptolysin O titers (ASOT) and anti-deoxyribonuclease B (anti-DNase B) will be measured at 0 months to establish upper limit of normal values and again at 6 months to compare across seasons. Anti-J8 antibodies will be measured at 0, 6 and 10 months and correlated with clinical disease and acquisition of GAS isolates. All GAS isolates from skin and throat swabs will undergo genetic sequencing of the N-terminal and C-repeat regions (for the J8 epitope) of the M protein at QIMR. One hundred fifty skin swabs and 150 throat swabs will undergo antimicrobial susceptibility testing against penicillin, erythromycin, clindamycin and chloramphenicol. The primary endpoints of the study are the incidence of culture confirmed GAS pharyngitis in 1000 children over 10 months and anti-J8 titers correlated against cases of pharyngitis and pyoderma in 600 children. The secondary endpoints of the study are: number of cases of pyoderma at 0,2,4,6,8,10 months; number of cases of scabies at 0,2,4,6,8,10 months; frequency of GAS isolation from throat swabs in 1000 asymptomatic children; proportion of children with pharyngitis who have clinical features suggestive of GAS pharyngitis; measurement of ASOT and anti-DNase B titres in 600 children - the upper limit of normal is defined at 80%; number of GAS isolates from throat swabs that contain the J8 epitope, and the overall emm-type distribution of GAS isolates; number of GAS isolates from skin swabs that contain the J8 epitope, and the overall emm-type distribution of GAS isolates; and antibiograms of GAS isolates from skin and throat to penicillin, clindamycin, erythromycin, and chloramphenicol.

ELIGIBILITY:
Inclusion Criteria:

* Informed consent will be obtained for all study participants.
* All children between 5-14 years of age are eligible for the study.

Exclusion Criteria:

None

Ages: 5 Years to 14 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 1000
Dates: Start 2006-01; Study Completion 2006-11

CONTACTS AND LOCATIONS:
Locations (1):
- Colonial War Memorial Hospital, Suva, Fiji